CLINICAL TRIAL: NCT03888417
Title: Tolerance of Therapeutic Plasma Exchange Performed in the Rennes University Hospital 2011-2018
Brief Title: TPE in Rennes Hospital
Acronym: COMPLASMA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3049_COMPLASMA
Record Dates: First submitted 2019-03-14; First posted 2019-03-25 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Therapeutic Plasma Exchange
Keywords: TPE; therapeutic plasma exchange; Side Effects
MeSH Terms: interventions — Plasma Exchange

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Therapeutic plasma exchange (TPE) — All TPEs were performed by the centrifugation technique using the Fresenius Kabi COMTEC machine

SUMMARY:
To assess the indications, tolerance and side effects of therapeutic plasma exchange (TPE) performed at a University Hospital over 8 years

DETAILED DESCRIPTION:
Indications were recorded from the patients electronic chart. Side effects were identified from the review of TPE monitoring forms completed prospectively by the nurse who performed the TPE during the course of the procedure

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who underwent TPE in Rennes University Hospital 2011-2018

Exclusion Criteria:

* Absence of the monitoring sheet during the EP session
* Refusal of patient participation after receipt of the information letter
* Persons over the age of majority who are subject to legal protection (protection of justice, guardianship, guardianship)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients who underwent TPE in Rennes University Hospital 2011-2018
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Frequency of side effects during Therapeutic plasma exchange | The inclusion day (retrospective study)
  Occurrence of side effects, regardless of their severity during therapeutic plasma exchange sessions (From start of care by the nurse including the preparation for the insertion of peripheral or central venous access to disconnection from the device and removal of peripheral lines or closing the CVC),. Main side effects recorded are hypotension, tachycardia, shock, anaphylaxis, seizure, cardiac arrest, respiratory failure, skin rash, urticaria, catheter dysfunction, catheter related infection hypocalcemia, alkalosis.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe CAMUS, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France

REFERENCES:
- [Derived] Coirier V, Lesouhaitier M, Reizine F, Painvin B, Quelven Q, Maamar A, Gacouin A, Tadie JM, Le Tulzo Y, Camus C. Tolerance and complications of therapeutic plasma exchange by centrifugation: A single center experience. J Clin Apher. 2022 Feb;37(1):54-64. doi: 10.1002/jca.21950. Epub 2021 Nov 17. PMID 34786746